CLINICAL TRIAL: NCT01779115
Title: Computerized Registry of Diabetes Patients in a Large Health Maintenance Organization in Israel
Brief Title: Registry of Diabetes Patients in a Large Health Maintenance Organization in Israel
Status: Enrolling by invitation | Type: Observational
Sponsor: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: MACCVREGDIAB
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Registry,Diabetes,Health Maintenance Organization
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A computerized registry of diabetes patients in a large health maintenance organization in Israel. The registry is aimed to be used by health professionals to identify diabetes patients and to follow the courses of their illnesses and risk factors.

DETAILED DESCRIPTION:
The registry was initiated in 1998 by Maccabi Healthcare services, which is the second largest publicly funded HMO in Israel,serving 24% of the total population with a nationwide distribution.

The registry uses advanced information technology that integrates personal computerized community and hospital records, data from laboratory tests, dispensed medications, physiological signals, radiological images, and reports from investigations and procedures.

ELIGIBILITY:
Inclusion Criteria:

Diabetic patient was defined according to the criteria suggested by American Diabetes Association - symptoms diagnosed as diabetes and fasting plasma glucose >125 mg/dl (7.0 lmol/l) or casual (namely, any time of day without regard to time since last meal) plasma glucose concentration P200 mg/dl. In order to reach maximal validity, we also included any patient who answered to one of the following: (1) purchased at least two hypoglycemic medications or single insulin dose during 6 months. (2) Had HbA1c result of at least 7.25%. HbA1c of 6.5% was used as entry criterion to registry only when the patient was diagnosed as diabetic.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes patients.
Sampling Method: Non-Probability Sample
Enrollment: 126000 (Estimated)
Dates: Start 1998-01; Primary Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence rates of Diabetes | Up to 100 years

SECONDARY OUTCOMES:
Rates of performance of eye examinations,blood and urine tests | up to 100 years
Number and types of Drugs purchased | 100 years
Number of visits to physician offices | up to 100 years

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chodick, PHD, Study Director — Head,Epidemiology & Database Reseaech Unit, Medical Division, Maccabi H.S
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel

REFERENCES:
- [Result] Chodick G, Heymann AD, Shalev V, Kookia E. The epidemiology of diabetes in a large Israeli HMO. Eur J Epidemiol. 2003;18(12):1143-6. doi: 10.1023/b:ejep.0000006635.36802.c8. PMID 14758871
- [Result] Heymann AD, Chodick G, Halkin H, Karasik A, Shalev V, Shemer J, Kokia E. The implementation of managed care for diabetes using medical informatics in a large Preferred Provider Organization. Diabetes Res Clin Pract. 2006 Mar;71(3):290-8. doi: 10.1016/j.diabres.2005.07.002. Epub 2005 Aug 19. PMID 16112245